CLINICAL TRIAL: NCT06213844
Title: A Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of IBI3002 in Healthy Participants and Participants With Mild to Moderate Asthma
Brief Title: A First-in-human, Single-ascending-dose Study of IBI3002 in Healthy Participants and Mild to Moderate Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3002A101AU
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants; Asthma
MeSH Terms: conditions — Asthma | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of Placebo administered subcutaneously on Day 1
  Interventions: Drug: Placebo
- IBI3002 (Experimental): Single dose of IBI3002 (Dosage 1, Dosage 2, Dosage 3, Dosage 4, Dosage 5, Dosage 6) administered subcutaneously on Day 1
  Interventions: Drug: IBI3002

INTERVENTIONS:
Drug: IBI3002 — Single dose of IBI3002 (Dosage 1, Dosage 2, Dosage 3, Dosage 4, Dosage 5, Dosage 6), administered subcutaneously on Day 1
  Other Names: ICS, alone or in combination with LABA
  Arms: IBI3002
Drug: Placebo — Single dose of Placebo, administered subcutaneously on Day 1
  Other Names: ICS, alone or in combination with LABA
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, phase 1, single-ascending-dose study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of IBI3002 in healthy participants and mild to moderate asthmatics. Subjects will be randomly assigned to different dosages of IBI3002 and matched placebo groups. The entire trial cycle includes a 4-week screening period, 1-day treatment period and 5-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign an Institutional Review Board (IRB) approved informed consent form before any study specific procedures.
2. Participants must be between 18 and 55 years old, inclusive.
3. Participants must have a body mass index (BMI) between 18 to 32 kg/m2, inclusive.
4. Participants of childbearing potential and their partners should use highly effective methods of birth control during the study and until 6 months after the study.
5. Participants with asthma must have:

   * Documented physician diagnosis of asthma for at least 12 months prior to screening and confirmed by the investigator;
   * Elevated FeNO defined as ≥ 25ppb;
   * Documented and stable GINA 2023 recommended Step 1~3 controller treatment (defined as ≤ 250μg fluticasone propionate dry powder formulation equivalent total daily dose of ICS, alone or in combination with LABA) for the last 3 months prior to screening;
   * Pre-BD FEV1 ≥ 60% of prediction and Post-BD FEV1/forced vital capacity (FVC) > 70%.

Exclusion Criteria:

1. History of allergies to any components of IBI3002 or placebo.
2. History of blood or needle sickness, or those who cannot tolerate venipuncture.
3. Female participants who are pregnant or breastfeeding at screening or randomization.
4. History of participating in a clinical trial within 1 month or 5 half-lives of the test drug (whichever is longer) prior to randomization, or those who are currently participating in a clinical trial.
5. History of severe infection or significant injury within 6 months, or surgery within 3 months, or any infection requiring systemic medication within 1 month prior to screening or randomization.
6. History of live or attenuated vaccination within 1 month prior to randomization, or those who plan to be vaccinated during the study.
7. For asthmatics only: history of a life-threatening asthma attack that required mechanical ventilation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years prior to randomization.
8. For asthmatics only: history of asthma worsen or exacerbation resulting in emergency room (ER) visits or overnight hospitalizations, or an increase in asthma maintenance therapy, or use of systemic glucocorticoids within the last 3 months prior to randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with AEs/SAEs | Baseline up to Day 36
  Incidence of adverse events and severe adverse events

SECONDARY OUTCOMES:
PK parameter: Cmax | Baseline up to Day 36
  Observed maximum plasma concentration
PK parameter: tmax | Baseline up to Day 36
  Time to achieve Cmax
PK parameter: AUC | Baseline up to Day 36
  Area under the plasma concentration-time curve
Immunogenicity profiles | Baseline up to Day 36
  Frequency and titers of anti-drug antibody (ADA)
PD profile (only in asthmatics): TARC (CCL17) | Baseline up to Day 36
  Change from baseline in peripheral blood TARC (CCL17) level
PD profile (only in asthmatics): IL-13 | Baseline up to Day 36
  Change from baseline in peripheral blood IL-13 level
PD profile (only in asthmatics): IgE | Baseline up to Day 36
  Change from baseline in peripheral blood Immunoglobulin
PD profile (only in asthmatics): Eosinophil | Baseline up to Day 36
  Change from baseline in peripheral blood eosinophil level
Clinical profile (only in asthmatics): FeNO | Baseline up to Day 36
  Change from baseline in Fractional exhaled Nitric Oxide
Clinical profile (only in asthmatics): Spirometry | Baseline up to Day 36
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second (Pre-BD FEV1)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No